CLINICAL TRIAL: NCT06431191
Title: Does Medial Raw Anchor Necessary During Tendon Repair Combined With Microfracture in Small to Medium Size Rotator Cuff Tear
Brief Title: Does Medial Raw Anchor Necessary During Tendon Repair Combined With Microfracture
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Jishuitan Hospital (Other)
Responsible Party: Principal Investigator, Yi Lu, Director of Sports Medicine Service of Beijing Jishuitan hospital, Beijing Jishuitan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: luyi
Record Dates: First submitted 2023-03-18; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Full Rotator Cuff Tear; Microfracture Procedure; Double Raw Repair; Lateral Raw Repair

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): lateral raw repair for full tear rotator cuff combined microfracture procedure
  Interventions: Procedure: lateral raw
- Control group (Placebo Comparator): double raw repair for full tear rotator cuff combined microfracture procedure
  Interventions: Procedure: double raw

INTERVENTIONS:
Procedure: lateral raw — lateral raw repair for full tear rotator cuff combined microfracture procedure, without medial raw
  Arms: Study group
Procedure: double raw — double raw repair for full tear rotator cuff combined microfracture procedure
  Arms: Control group

SUMMARY:
This study is a prospective randomized controlled study of rotator cuff repair with lateral raw or double raw combined with microfracture procedure. The patients with rotator cuff tear were randomly divided into groups before the operation. The patients were followed up before and, 3 months, 6 months, 12 months and 24 months after surgery. In different time periods, the quantitative and qualitative indicators including pain, functional score, muscle strength, MRI performance, etc. were compared between groups at the same time period to evaluate the difference in the effect of double raw or only lateral raw repair combined with microfracture on the treatment of rotator cuff. In order to figure out whether medial raw anchor necessary during tendon repair combined with microfracture in small to medium size rotator cuff tear.

ELIGIBILITY:
Inclusion Criteria:

* Arthroscopy confirmed small to medium full rotator cuff tear
* Unilateral rotator cuff injury
* Voluntarily accept randomized controlled grouping, cooperate with treatment and follow up patients
* Young and middle-aged patients aged 20 to 60

Exclusion Criteria:

* Previous shoulder surgery (incision or arthroscopy)
* Combined with diseases of other parts of the same limb
* Combined with Bankart injury, acromioclavicular joint disease, greater tuberosity fracture, glenoid fracture and so on
* Bilateral onset
* Unable or unwilling to receive clinical follow-up

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
rotator cuff re-tear rate | 6, 12, 24 months postoperatively
  the rotator cuff re-tear rate was measured by MRI, MRI was performed to identify the status of the tendon

SECONDARY OUTCOMES:
VAS (Visual Analogue Scale) | 1,2,3,7 days postoperatively and 3,6,12,24 months postoperatively
  A score used to evaluate the pain, higher scores mean a worse outcome.
ASES(American Shoulder and Elbow Surgeons'Form) | 3,6,12,24 months postoperatively
  A score used to evaluate the shoulder function, higher scores mean a better outcome.
Constant score | 3,6,12,24 months postoperatively
  A score used to evaluate the shoulder function,higher scores mean a better outcome.
UCLA (University LosAngeles scoring system) | 3,6,12,24 months postoperatively
  A score used to evaluate the shoulder function
SST (simple shoulder test) | 3,6,12,24 months postoperatively
  A score used to evaluate the shoulder function,higher scores mean a better
front extension, external rotation and internal rotation strength of shoulder | 6,12,24 months postoperatively
  Use a dynamometer to measure in N
surgical time | immediately after the surgery
  surgical time, describe with minute
Hospitalization expenses | immediately after the patient discharge
  payment during the hospital stay, Treatment fee is calculated in RMB

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Jishuitan hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No